CLINICAL TRIAL: NCT04949360
Title: Evaluation of SleepUp Digital CBTi-based Platform in the Treatment of Insomnia
Brief Title: SleepUp Digital CBTi-based Platform for Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SleepUp Tecnologia em Saúde Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SleepUp_#01; 34113520.1.0000.5494 (Other: Brazilian National Comission of Research Ethics)
Record Dates: First submitted 2021-06-13; First posted 2021-07-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Sleep Disorder; Sleep Hygiene
Keywords: Insomnia; Sleep; Cognitive-behavioral therapy; CBTi
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Sleep Hygiene | interventions — Complementary Therapies

STUDY DESIGN:
Intervention Model Description: Phase 1=Participants will be randomized and distributed in four parallel and independent groups.
  Phase 2=Participants will be randomized and distributed in three parallel and independent groups.
Who Masked: Outcomes Assessor
Masking Description: The participants cannot be blinded considering the type of intervention being tested. The allocation codes will be concealed and only three members of the research team will have access to the codes and randomization table. All the outcomes will be either collected automatically (via software) or by hired professionals unaware of the objectives of this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (4):
- Standard CBTi (CBTi-S): (Active Comparator): This is a positive control group/active comparator, in which standard CBTi (the golden standard behavioral treatment for insomnia) will be made available. This treatment consists of an eight-week treatment composed by weekly and structured appointments with a board-certified sleep psychologist. The professionals performing the CBTi sessions will not be part of the research team. The appointments will be made remotely (video calls with psychologists), which have already been proven to be equivalent to the in-person CBTi.
  Interventions: Behavioral: Regular Cognitive Behavioural Therapy for Insomnia
- Minimal intervention - Sleep hygiene (MI-SH): (Placebo Comparator): This group corresponds to a negative control group/placebo comparator, subjected to minimal intervention. It is based on the delivery of informative material regarding normal sleep pattern and sleep hygiene (through SleepUp app). This procedure is more adequate as a control than the commonly used no-treatment or waiting list controls, due to the behavioral nature of insomnia.
  Interventions: Behavioral: Sleep hygiene - minimal intervention
- Online CBTI (CBTI-O) (Experimental): This group will receive access to an eight-week CBTi-based treatment through the SleepUp app. The platform will be updated into a non-commercial version, and all features other than the CBTi track will be removed. This way, the participants of this group will receive interventions equivalent to the standard in-person CBTi, but provided through a digital platform.
  Interventions: Behavioral: Online Cognitive-Behavioral Therapy for Insomnia and complementary therapies
- Online CBTi + additional features (CBTi-O+) (Experimental): This group will have access to the complete premium version of SleepUp platform. It includes those presented in the CBTi-O group and other therapeutic and complementary features (including meditation audios and videos, mindfulness therapy, relaxation soundtracks, sleep hygiene tips, virtual assistant, and telehealth.
  Interventions: Behavioral: Online Cognitive-Behavioral Therapy for Insomnia and complementary therapies

INTERVENTIONS:
Behavioral: Online Cognitive-Behavioral Therapy for Insomnia and complementary therapies — The CBTi-O and CBTi-O+ interventions are based on real life user experience. The users will have access to different versions of the platform. The intervention will last eitght weeks.
  Arms: Online CBTI (CBTI-O); Online CBTi + additional features (CBTi-O+)
Behavioral: Regular Cognitive Behavioural Therapy for Insomnia — This is the gold standard behavioral treatment for insomnia and will be performed by independent board-certified sleep psychologists. The treatments will last eight weeks and the appointments will be made by video-calls.
  Arms: Standard CBTi (CBTi-S):
Behavioral: Sleep hygiene - minimal intervention — It is composed by educational material about normal sleep pattern and sleep hygiene. It will be delivered by SleepUp app.
  Arms: Minimal intervention - Sleep hygiene (MI-SH):

SUMMARY:
Cognitive-Behavioral Therapy for insomnia (CBTi) is a well-established therapeutic intervention for insomnia. SleepUp provides a digital therapeutics platform based on CBTi and additional features. This clinical trial aims at analyzing the efficacy of the CBTi-based platform offered by SleepUp in reducing symptoms of insomnia and will be conducted in 2 phases.

Phase 1

The sample will be composed of 160 individuals, both males and females, from 20 to 60 years old, with insomnia symptoms considered as at least mild. Those who accept to participate will be randomized and distributed in four groups:

* Standard CBTi (CBTi-S): This treatment consists of an eight-week treatment composed by weekly and structure appointments with board-certified sleep psychologists. The appointments will be made remotely (video calls with psychologists).
* Minimal intervention - Sleep hygiene (MI-SH): This group will receive an educational program on sleep hygiene through the SleepUp app. Its content covers topics that are also covered in the online CBTi sessions. This procedure is more adequate as a control than the commonly used no treatment or waiting list controls, due to the behavioral
* Online CBTI (CBTI-O): This group will receive access to an eight-weeks CBTi-based treatment through the SleepUp app. The participants of this group will receive interventions equivalent to the standard in-person CBTi, but provided through a digital platform.
* Online CBTi + additional features (CBTi-O+): This group will have access to the complete premium version of SleepUp platform. It includes those presented in the CBTi-O group and other therapeutic and complementary features (including meditation audios and videos, mindfulness therapy, relaxation soundtracks, sleep hygiene tips, virtual assistant, and telehealth.

All participants in all groups will be assessed periodically throughout the eight weeks of intervention with standard sleep questionnaires and sleep logs. Equivalent intervals will be applied to the MI-SH group.

Phase 2

This phase will comprise 120 individuals, both males and females, from 20 to 60 years old, with insomnia symptoms considered as at least mild. Those who accept to participate will be randomized and distributed in three groups:

* Minimal intervention - Sleep hygiene (MI-SH): This group will receive an educational program on sleep hygiene through the SleepUp app. Its content covers topics that are also covered in the online CBTi sessions. This procedure is more adequate as a control than the commonly used no treatment or waiting list controls, due to the behavioral
* Online CBTI (CBTI-O): This group will receive access to an eight-weeks CBTi-based treatment through the SleepUp app. The participants of this group will receive interventions equivalent to the standard in-person CBTi, but provided through a digital platform.
* Online CBTi + additional features (CBTi-O+): This group will have access to the complete premium version of SleepUp platform. It includes those presented in the CBTi-O group and other therapeutic and complementary features (including meditation audios and videos, mindfulness therapy, relaxation soundtracks, sleep hygiene tips, virtual assistant, and telehealth.

All participants in all groups will be assessed periodically throughout the eight weeks of intervention with standard sleep questionnaires and sleep logs. Equivalent intervals will be applied to the MI-SH group.

DETAILED DESCRIPTION:
Cognitive-Behavioral Therapy for insomnia (CBTi) is a well-established therapeutic intervention for insomnia. In its standard presentation, it is composed by 6 to 12 weekly appointments with a board-certified sleep psychologist. SleepUp provides a digital therapeutics platform based on CBTi and additional features. This clinical trial aims at analyzing the efficacy of the CBTi-based platform offered by SleepUp in reducing symptoms of insomnia.

The participants will be recruited based on advertising on social media and invited to participate. Those participants who are eligible in accordance to the inclusion and exclusion criteria will be contact by a member of the research team who will provide a consent form and will explain the terms and conditions of this research project. The sample will be composed of 160 individuals in Phase 1 and by 120 individuals in Phase 2, both males and females, from 20 to 60 years old, with insomnia symptoms considered as at least mild, according to the Insomnia Severity Index (ISI). All groups shall have similar proportions of gender and of insomnia symptoms severity.

Phase 1

Those who accepted to participate will be randomized and distributed in four groups:

* Standard CBTi (CBTi-S): This is a positive control group, in which standard CBTi (the golden standard behavioral treatment for insomnia) will be made available. This treatment consists of an eight-week treatment composed by weekly and structure appointments with psychologists. Only psychologists board-certified in sleep medicine will perform the CBTi sessions, and none of them are part of the research team. The appointments will be made remotely (video calls with psychologists), which have already been proven to be equivalent to the in-person CBTi.
* Minimal intervention - Sleep hygiene (MI-SH): This group corresponds to a negative control group, subjected to minimal intervention. It is based on the delivery of informative material regarding normal sleep pattern and sleep hygiene (through SleepUp app). This procedure is more adequate as a control than the commonly used no treatment or waiting list controls, due to the behavioral nature of insomnia.
* Online CBTI (CBTI-O): This group will receive access to an eight-week CBTi-based treatment through the SleepUp app. The platform will be updated into a non-commercial version. This way, the participants of this group will receive interventions equivalent to the standard in-person CBTi, but provided through a digital platform.
* Online CBTi + additional features (CBTi-O+): This group will have access to the complete premium version of SleepUp platform. It includes those presented in the CBTi-O group and other therapeutic and complementary features (including meditation audios and videos, mindfulness therapy, relaxation soundtracks, sleep hygiene tips, virtual assistant, and telehealth.

Phase 2

Those who accepted to participate will be randomized and distributed in three groups:

* Minimal intervention - Sleep hygiene (MI-SH): This group corresponds to a negative control group, subjected to minimal intervention. It is based on the delivery of informative material regarding normal sleep pattern and sleep hygiene (through SleepUp app). This procedure is more adequate as a control than the commonly used no treatment or waiting list controls, due to the behavioral nature of insomnia.
* Online CBTI (CBTI-O): This group will receive access to an eight-week CBTi-based treatment through the SleepUp app. The platform will be updated into a non-commercial version. This way, the participants of this group will receive interventions equivalent to the standard in-person CBTi, but provided through a digital platform.
* Online CBTi + additional features (CBTi-O+): This group will have access to the complete premium version of SleepUp platform. It includes those presented in the CBTi-O group and other therapeutic and complementary features (including meditation audios and videos, mindfulness therapy, relaxation soundtracks, sleep hygiene tips, virtual assistant, and telehealth.

All participants in all groups will be assessed periodically throughout the eight weeks of intervention. Equivalent intervals will be applied to the SH-MI group. The following clinical questionnaires and scales will be used:

* Sleep log: It includes self-reported items regarding wake and bedtime, sleep latency and other sleeping habits. It allows the calculation of total sleep time, sleep efficiency and wake time after sleep onset. Fille daily.
* Morningness and Eveningness Questionnaire: It evaluates chronotype based on 19 items, allowing categorizing the participants according to the following categories: morning type (definitive or moderate), intermediate, or evening type (definitive or moderate). Applied once, in the first week of follow up.
* Insomnia Severity Index: It evaluates the presence and severity of insomnia, categorizing the participants according to the following categories: no, mild, moderate or severe insomnia. Applied once every two weeks.
* Epworth Sleepiness Scale: It evaluates excessive daytime sleepiness by inquiring about the chance of sleeping in eight daily situations. Scores higher than 10 indicates excessive daytime sleepiness. Applied once every two weeks.
* Pittsburgh Sleep Quality Index: It evaluates overall sleep quality based on 19 self-reported items. Scores higher than 5 indicates poor sleep quality. Applied once every two weeks.
* Sleep Hygiene Index: It habits related to sleep hygiene, based on 13 self-reported items.

ELIGIBILITY:
Inclusion Criteria:

* Literate Brazilian portuguese speakers.
* Insomnia symptoms (as measured by ISI).
* An Android-based smartphone or tablet with access to the Internet.

Exclusion Criteria:

* Previous experience with CBTi.
* Use of sleeping pills or any other treatment for insomnia for two or more days a week in the last three months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to the treatment | From enrollment (baseline) to the end of treatment at 8 weeks
  It will be measured as the percentage of participants who completed the treatment, out of those who effectively initiated it. Dropouts will be considered whenever a participants fail to comply with the tasks relative to each group for two consecutive weeks, or postpone the completion of these tasks for three times. These tasks refer to the responses to periodic questionnaires and to the completion of the CBTi or CBTi-O sessions (when applicable).The aim of this comparison is to evaluate whether the adherence rate in the CBTi-O and CBTi-O+ groups are similar to the standard treatment (CBTi-S) or higher than the minimal treatment (MI-SH).
Response to treatment | From enrollment (baseline) to the end of treatment at 8 weeks
  Patients are considered to be responsive to treatment if the ISI score is at least 7 points lower than on the basal evaluation.
Remission of symptoms | From enrollment (baseline) to the end of treatment at 8 weeks
  Patients are considered to be with no symptoms of insomnia if the ISI score is lower then 8.

SECONDARY OUTCOMES:
Self-reported sleep efficiency | From enrollment (baseline) to the end of treatment at 8 weeks
  Sleep efficiency will be measured by sleep logs
Sleep hygiene | From enrollment (baseline) to the end of treatment at 8 weeks
  Sleep hygiene habits will be measured by the Sleep Hygiene Index
Excessive daytime sleepiness | From enrollment (baseline) to the end of treatment at 8 weeks
  Excessive daytime sleepiness will be measured using the Epworth Sleepiness Scale
Sleep quality | From enrollment (baseline) to the end of treatment at 8 weeks
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index
Self-reported sleep latency | From enrollment (baseline) to the end of treatment at 8 weeks
  Sleep latency will be measured by sleep logs
Self-reported sleep duration | From enrollment (baseline) to the end of treatment at 8 weeks
  Sleep duration will be measured by sleep logs

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel N. Pires, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- SleepUp Tecnologia em Saúde LTDA, São Caetano do Sul, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The dissemination of Individual Participant Data (IPD) from this study is strictly limited by restrictions on the release of intellectual property, concerns regarding participant privacy and confidentiality, and the absence of explicit consent for extensive data sharing. However, upon reasonable request and subject to approval by the study's principal investigator, anonymized datasets may be provided to qualified researchers. It is imperative that requests include a thorough research proposal and a rationale that substantiates the need for the resources in question.